CLINICAL TRIAL: NCT04056169
Title: Comparison of High-dose Rosuvastatin Versus Low-dose Rosuvastatin Plus Ezetimibe on Carotid Plaque Inflammation in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: seeCAP
Record Dates: First submitted 2019-08-08; First posted 2019-08-14 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Acute Coronary Syndrome; Carotid Atherosclerotic Plaque With Inflammation
Keywords: rosuvastatin; ezetimibe/rosuvastatin; carotid plaque inflammation; fluorodeoxyglucose F18; positron emission tomography
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin (Active Comparator): rosuvastatin 20 mg once a day for 6 months
  Interventions: Drug: high-dose rosuvastatin
- ezetimibe/rosuvastatin (Experimental): ezetimibe/rosuvastatin 10/5 mg once a day for 6 months
  Interventions: Drug: low-dose rosuvastatin plus ezetimibe

INTERVENTIONS:
Drug: high-dose rosuvastatin — rosuvastatin 20 mg once a day for 6 months
  Arms: Rosuvastatin
Drug: low-dose rosuvastatin plus ezetimibe — ezetimibe/rosuvastatin 10/5 mg once a day for 6 months
  Arms: ezetimibe/rosuvastatin

SUMMARY:
Combination therapy of ezetimibe with a low-dose statin is occasionally used to avoid statin-related side effects in clinical practice among patients with atherosclerotic cardiovascular disease. This approach is equivalent to high-dose statin therapy to decrease LDL cholesterol level by >50%, allowing such patients to achieve LDL cholesterol target. However, it remains uncertain whether combination therapy with ezetimibe and low-dose statin verse high-dose statin monotherapy similarily suppress atherosclerotic plaque inflammation. This study is to compare high-dose rosuvastatin versus low-dose rosuvastatin plus ezetimibe on carotid plaque inflammation in patients with acute coronary syndrome using 18F-fluorodeoxyglucose (18FDG) positron emission tomography (PET) imaging.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 19 years
2. acute coronary syndrome, carotid artery disease (diameter stenosis 20-50%), and at least one 18FDG uptake lesion in the carotid artery (target to background ratio (TBR) ≥ 1.6) by 18FDG PET/CT imaging
3. written consent

Exclusion Criteria:

1. previous history of carotid endarterectomy or stenting
2. schedule for cardiac or major surgery within the next 6 months
3. statin or ezetimibe therapy in the past 4 weeks
4. chronic disease needed to be treated with oral, intravenous, or intraarticular steroid
5. end-stage renal disease
6. chronic liver disease
7. history of cancers within the past 3 years
8. pregnant, breast-feeding or child-bearing potential
9. expected life expectancy within 2 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Percent change in most-diseased segment (MDS)-tissue blood ratio (TBR) of the index vessel | 6 months

SECONDARY OUTCOMES:
Change in MDS TBR | 6 months
Change in whole vessel TBR within the index vessel | 6 months
Change in whole vessel TBR of the aorta | 6 months
Change in total cholesterol | 6 months
Change in triglyceride | 6 months
Change in HDL-cholesterol | 6 months
Change in LDL-cholesterol | 6 months
Change in high sensitive C-reactive protein | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul